CLINICAL TRIAL: NCT01668108
Title: Open, Multicenter Observational Study of Paclitaxel Utilized in Mono- or Combination Therapy for the Treatment of Breast Cancer, Non-small Cell Lung Cancer and Ovarial Cancer.
Brief Title: A Non Interventional Study With Paclitaxel Onkovis (Paclitaxel) Utilized for the Treatment of Cancer
Status: Completed | Type: Observational
Sponsor: Onkovis GmbH (Industry)
Collaborators: AKP Freiburg GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ONKOPAC 01
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma
Keywords: carcinoma; breast cancer; non-small cell lung cancer; ovarial cancer; ambulant chemotherapy; treatment cycles; Paclitaxel; Paclitaxel onkovis; Quantity of Paclitaxel; Packaging Sizes
MeSH Terms: conditions — Carcinoma; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- carcinoma, Paclitaxel onkovis (Paclitaxel): treatment in mono- or combination therapy with Paclitaxel of breast-, non-small cell lung- and ovarial cancer.

SUMMARY:
The main purpose of this observational study with Paclitaxel is to determine the number of treatment cycles and the quantity of Paclitaxel onkovis needed therefore under the special circumstance of ambulant chemotherapy.

onkovis aims an economical utilization of the chemotherapeutics.The provision with adapted packaging sizes as to decrease the excess quantity to be discarded follows also this objective.

Secondary objectives are the survey of the side effects of Paclitaxel onkovis in comparison to Docetaxel. To this purpose, data regarding co medications and adverse events are also collected.

ELIGIBILITY:
Inclusion Criteria:

* Indication for Paclitaxel according to the SmPC and treating physician

Exclusion Criteria:

* according to the Paclitaxel SmPC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated in practices, clinics, hospitals
Sampling Method: Probability Sample
Enrollment: 770 (Actual)
Dates: Start 2012-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
the quantity of Paclitaxel onkovis needed pro treatment cycle | the time the participants will be followed depends on the number of treatment cycles; that means the time frame may extend up to 24 weeks (8 cycles).
  Determine the quantity of Paclitaxel onkovis needed pro treatment cycle

SECONDARY OUTCOMES:
adverse events during and after treatment in comparison to Docetaxel onkovis | up to 24 weeks (8 cycles)
  The number and kind of adverse events during and after the intra-venous application of Paclitaxel will be assessed, documented and compared to those of Docetaxel.

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Practice, Brandenburg
  - Practice, Chemnitz
  - Practice, Dresden
  - Practice, Mühlhausen
  - Practice, Plauen